CLINICAL TRIAL: NCT03269058
Title: Effects of Dapagliflozin on Lipoprotein Kinetics in Patients With Type 2 Diabetes
Brief Title: Evaluate the Effects of Dapagliflozin in Patients With Type 2 Diabetes
Acronym: Cinétique DAPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VERGES AZ 2015
Record Dates: First submitted 2017-08-25; First posted 2017-08-31 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Type-2 Diabetes; Oral Antidiabetics
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients not treated with statins (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Placebos
- Patients treated with statins (Experimental)
  Interventions: Drug: Dapagliflozin; Drug: Placebos

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg daily per os
Drug: Placebos — Placebo of Dapagliflozin per day per os

SUMMARY:
This study will make it possible to better understand the mechanisms responsible for the increase in bad cholesterol levels observed in patients with type 2 diabetes treated with Dapagliflozin, an antidiabetic treatment made by Astrazeneca.

The information will:

* reveal what is not working properly
* make it possible to choose the most appropriate treatments against cholesterol to compensate for this impaired functioning

This biomedical research will take place at the University Hospitals of DIJON and NANTES.

* 28 patients will take part: 20 patients will be given Dapagliflozin and 8 patients will be given the placebo.
* The study treatment will be randomised: patients will be given either Dapagliflozin or the placebo. The treatment duration is 6 months.
* Moreover, during the inclusion visit and at the end of the study (6 months after the start of treatment), a kinetics study, to follow the production and elimination of cholesterol, will be conducted. This will involve administering amino acids that have been specifically synthesised for this purpose.
* Participation in the study will last 6 months and include 4 protocol visits.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written consent
* type 2 diabetes treated with OAD (metformin and/or sulfonylurea and/or glinides and/or acarbose and/or DPPIV inhibitors)
* Stable treatment for 3 months
* HbA1c between 7.5% and 10%
* Age between 30 and 65 years
* BMI between 25 and 35 kg/m²
* Triglycerides < 300 mg/dl
* Half of the patients being treated with statins
* eGFR > 75 ml/min/1.73 m² at inclusion

Exclusion Criteria:

* persons without national health insurance cover
* patients treated with Insulin or a GLP-1 agonist
* Patients under guardianship
* patients treated with lipid-lowering drugs (except statins for 50% of patients)
* kidney failure
* liver failure or abnormal liver function ASAT or ALAT >3 x upper limit of normal
* total bilirubin >2mg/dl
* intestinal disease
* serological evidence of an active liver infection (surface antigen of hepatitis B, hepatitis C antibodies, hepatitis B IgM antibodies)
* Pregnancy, breastfeeding
* hypersensitivity to the active substance or to excipients
* patients with volume depletion, for example due to an acute disease (gastro-intestinal disease)
* patients treated with loop diuretics or thiazides

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline the rate of production of VLDL Apo B | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the rate of production of IDL Apo B | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the rate of production of LDL Apo B | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the rate of production of HDL Apo A1 | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the Fractional Catabolic Rate of VLDL1 Apo B | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the Fractional Catabolic Rate of VLDL2 Apo B | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the Fractional Catabolic Rate of IDL Apo B | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the Fractional Catabolic Rate of LDL Apo B | 15 days before treatment initiation, Day 0, Day 90 and Day 180
Change from baseline the Fractional Catabolic Rate of HDL 'Apo A1 | 15 days before treatment initiation, Day 0, Day 90 and Day 180

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Dijon Bourgogne, Dijon
  - CHU de Nantes, Nantes